CLINICAL TRIAL: NCT01192958
Title: A Study to Validate a New Oral Fluid/Saliva Antibody Test for Novel H1N1v Influenza
Acronym: Snuffles
Status: Completed | Type: Observational
Sponsor: Public Health England (Other Government)
Responsible Party: Professor Liz Miller, Health Protection Agency
Other Study IDs: OFLU
Record Dates: First submitted 2010-08-31; First posted 2010-09-01 (Estimated); Last update posted 2010-09-01 (Estimated); Status verified 2009-12

CONDITIONS: H1N1 Virus
Keywords: swine flu; novel h1n1v; novel h1n1; h1n1
MeSH Terms: conditions — Orthomyxoviridae Infections

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

SUMMARY:
At present influenza immunity can only be reliably confirmed by a blood test. This test is invasive for the patient. This study is intended to validate an oral fluid/saliva antibody test for the variant Swine Influenza H1N1. If such a test were available, this painless and non invasive test will improve direct clinical care to an individual as well as significantly help guide future public health management of the pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Participants of the clinical service evaluation of novel H1N1v vaccine
* First or second blood sample for the clinical service evaluation successfully collected

Exclusion Criteria:

* Withdrawn from clinical service evaluation of novel H1N1v vaccine
* Second blood sample for the clinical service evaluation not collected.

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects from primary care who are participating in the clinical service evaluation.
Sampling Method: Non-Probability Sample
Dates: Start 2010-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)